CLINICAL TRIAL: NCT02147210
Title: Chronic Transplant Glomerulopathy and Regulation of Expression of Ephrin B1
Acronym: GARRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 13 194 02; AOL 2013 (Other Grant/Funding Number: University Hospital Toulouse)
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Kidney Transplantation
Keywords: Chronic transplant glomerulopathy; antibody mediated rejection; Ephrin-B1
MeSH Terms: interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-Case: patients who developed CTG secondary to antibody-mediated kidney rejection (AMR), diagnosed by microscopic analysis.
  Interventions: Other: biological analysis
- 2-Control: patients with antibody-mediated kidney rejection (AMR) but without CTG
  Interventions: Other: biological analysis

INTERVENTIONS:
Other: biological analysis

SUMMARY:
The principal purpose is the study of the regulation of the expression of ephrin-B1 by immunofluorescence in kidney biopsies of patients with Chronic transplant glomerulopathy (CTG) compared to biopsies prior to the CTG, in same patients. Level of fluorescence in CTG biopsy will be the experimental reference value.

DETAILED DESCRIPTION:
Chronic transplant glomerulopathy (CTG) is a specific lesion of kidney transplantation and a poor prognostic factor affecting transplant survival. Diagnosis remains only microscopic and lesions are irreversible. Recent studies prove that there is a strong correlation between CTG and antibody mediated rejection (AMR) with a possible link with chronic aggression of the endothelial cell. However, for unknown reason, all AMR does not lead to a CTG. Our recent data on mice demonstrated that ephrin-B1 is expressed in the glomerular endothelial cells and knockout mice for the gene encoding ephrin-B1 develop progressively ultrastructural glomerular lesions close to modifications observed in CTG, as well as proteinuria and chronic renal failure, suggesting that ephrin B1 could participate to CTG. Moreover, in a preliminary study on human kidney transplant biopsy we observed decrease in ephrin-B1 immunofluorescence on glomerulus when CTG, even in low grade. These data, and ultrastructural modifications in Knock Out (KO) mice suggest that early regulation of kidney expression of ephrin-B1 in the glomerulus may occur during the process leading to the CTG as antibody-mediated kidney rejection (AMR).

The purpose of the study is to determinate if ephrin-B1 expression is modified in CTG.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patient for whom renal biopsies are stored in the "collection of the University Hospital Toulouse" (collection N° DC-2009-989) and who received information on the purpose of the study, use of biopsies and who has not manifested any opposition.
* Kidney transplant patient with iterative biopsies with at least: post-surgery biopsy D0 (or early post-transplant biopsy D7 and at least one biopsy protocol. - Age> 18 years Case group: - Kidney transplant patient, followed up by "organ transplant unity" of CHU Toulouse, with antecedent of CMR progressing to CTG between 2006 and 2013. Control group: - Kidney transplant patient, followed up by "organ transplant unity" of CHU Toulouse, with antecedent of CMR without progressing to CTG between 2006 and 2013

Exclusion Criteria:

* patient with uncontrolled hypertension - patient with diabetes mellitus -
* patient treated or who was treated with mTOR inhibitor - recurrence of the initial glomerular pathology - de novo glomerulopathy - patient including in another study with an exclusion period still going

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biopsies from patients corresponding to eligibility criteria (see below) will be selected from the list of kidney transplant patients followed up in the Toulouse University Hospital. They will be divided into two groups matched for age, sex and time of kidney transplantation (n = 30 for each group). Iterative biopsies are conserved in the collection of tissue samples of the CHU
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Expression level of ephrin-B1 in biopsies from kidney transplant | Day 1
  Analysis on all biopsies available from transplantation to Chronic transplant glomerulopathy by immunofluorescence (by anti-C4d)

SECONDARY OUTCOMES:
Level of expression of the gene encoding for ephrin-B1 | Day 1
  Analysis on all biopsies available from transplantation to Chronic transplant glomerulopathy by quantitative PCR (qPCR) and normalized to the expression of the gene encoding for GAPDH
Kinetics of expression of ephrin-B1 | Day 1
  Analysis on all biopsies available from transplantation to CTG by quantitative PCR (qPCR) and normalized to the expression of the gene encoding for GAPDH

CONTACTS AND LOCATIONS:
Overall Officials: Céline Guilbeau-Frugier, MD, Principal Investigator — Service d'Anatomie Pathologique et Histologie-Cytologie,Rangueil Hospital, University Hospital of Toulouse; Jean-Michel Senard, Md PhD, Study Director — Department of Pharmacology,Toulouse University Hospital and INSERM U1048
Locations (1):
- Service d'Anatomie Pathologique et Histologie-Cytologie Hôpital Rangueil, Toulouse, France